CLINICAL TRIAL: NCT07180810
Title: Effect of Low Dose Intravenous Dexmedetomidine on Post Anesthesia Discharge After Day Case Breast Cancer Surgery
Brief Title: Effect of Dexmedetomidine Infusion on Post Anesthesia Discharge Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-23-14
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2023-08

CONDITIONS: Post Anesthesia Discharge Time in Patients of Breast Cancer Surgery
Keywords: Breast cancer surgery, Dexmedetomidine, Post anesthesia discharge time

STUDY DESIGN:
Intervention Model Description: Group A being administered low dose intravenous dexmedetomidine infusion vs Group B being admissions IV normal saline infusion at rate 0.6mcg/kg/hour rate
Who Masked: Participant, Care Provider
Masking Description: Double blinded study, all participants, and the care provider providing anesthesia to the participants were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, receiving low dose dexmedetomidine infusion (Experimental): Group A, receiving low dose dexmedetomidine infusion at 0.6mcg/kg/hour rate
  Interventions: Drug: Dexmedetomidine infusion low dose
- Group B, receiving normal saline infusion as placebo (Placebo Comparator): normal saline being used as placebo at rate 0.6mch/kg/hour rate
  Interventions: Drug: Group B receiving normal saline

INTERVENTIONS:
Drug: Dexmedetomidine infusion low dose — low dose dexmedetomidine infusion at rate 0.6mcg/kg/hour rate .
  Arms: Group A, receiving low dose dexmedetomidine infusion
Drug: Group B receiving normal saline — Normal saline infusion at rate 0.6mcg/kr/hour rate
  Arms: Group B, receiving normal saline infusion as placebo

SUMMARY:
A randomised control trial evaluating the effect of low dose dexmedetomidine infusion on post anesthesia discharge time in patients of day case breast cancer surgery compared with placebo infusion. The primary outcome was to compare the frequency of early discharge in each group.

DETAILED DESCRIPTION:
A prospective Randomised control trial evaluating the effect of low dose dexmedetomidine infusion on post anesthesia discharge time in patients of day case breast cancer surgery compared with placebo infusion. The primary outcome was to compare the frequency of early discharge in each group. Early discharge was defined as within two hours. The sample size was of 82 female patients with a specific inclusion and exclusion criteria. Randomisation was done through computer software and the trial was double blinded. SPSS version 22 will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 yrs, ASA 1 and 2, elective breast cancer surgery

Exclusion Criteria:

* BMI greater than 35, CKD stage 3 or greater, known drug allergy to study drug, bradycardia, history of PONV, patients on antiepileptics

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 82 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Frequency of early discharge | 120 minutes
  post anesthesia discharge time within 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Almas nil Iqbal, FRCA, Study Chair — Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore, Pubjab, Pakistan

IPD SHARING:
Plan to Share IPD: No
undecided

REFERENCES:
- See also: Reference study from which sample size was calculated — https://journals.lww.com/ijaweb/fulltext/2018/62030/Role_of_dexmedetomidine_as_an_anaesthetic_adjuvant.5.aspx